CLINICAL TRIAL: NCT02521623
Title: SurgiMend® vs. Strattice™ in Direct to Implant Breast Reconstruction- A Prospective Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Alexander Juhl Andersen, MD, Ph.D.-student, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 48607
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Breast Neoplasms
Keywords: Acelullar Dermal Matrix; Immediate Breast Reconstruction; Breast Implant
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgimend (Experimental): Patients randomized to this arm will receive SurgiMend® Acellular Dermal Matrix in their direct to implant primary breast reconstruction.
  Interventions: Device: SurgiMend® Acellular Dermal Matrix
- Strattice (Active Comparator): Patients randomized to this arm will receive Strattice™ Acellular Dermal Matrix in their direct to implant primary breast reconstruction.
  Interventions: Device: Strattice™ Acellular Dermal Matrix

INTERVENTIONS:
Device: SurgiMend® Acellular Dermal Matrix — See arm description.
  Arms: Surgimend
Device: Strattice™ Acellular Dermal Matrix — See arm description.
  Arms: Strattice

SUMMARY:
An increasing number of women undergo an immediate breast reconstruction, where the mastectomy and the breast reconstruction are performed in the same surgery. To aid survival of the mastectomy skin flaps, and to provide better aesthetic results acellular dermal matrixes (ADMs) are used to reinforce the breast. There are several different types of ADM available for this purpose. In this randomized clinical trial, the following study will investigate two different types of ADM (Strattice™ and SurgiMend®) in an immediate breast reconstructive setting. Sixty patients will be allocated on a 1:1 ratio to receive either Strattice™ or SurgiMend® ADM. Patients scheduled for immediate breast reconstruction with ADM at pt. of Plastic and Reconstructive Surgery at Aarhus University Hospital, Aarhus, Denmark will be offered participation. In total, 60 patients will be included. Outcome parameters of interest are complication rate, patient satisfaction, aesthetic result and cost of the procedure. Satisfaction and aesthetic result will be measured at 4 and 12 months post surgery.

DETAILED DESCRIPTION:
Introduction

An increasing number of Danish women undergo genetic counseling for hereditary breast cancer. If the patient´s lifetime risk is evaluated to be more than 30%, the patient may choose to undergo a risk-reducing mastectomy (prophylactic mastectomy) to reduce the risk of developing breast cancer. The mastectomy is mostly performed as a skin-sparing procedure, where only the nipple area and the breast tissue is removed leaving the skin envelope intact, in order to preserve the breast skin for an immediate breast reconstruction. In select cases the surgery may be performed as a nipple-sparing procedure. Additionally, there is an increasing group of women diagnosed with multifocal DCIS who choose risk-reducing mastectomy with an immediate reconstruction.

In order for the risk-reducing mastectomy to be effective, it is of utmost importance that all the breast tissue is removed. This leaves the skin flaps covering the breast thin and vulnerable to necrosis, if not handled with utmost care. In order to spare the mastectomy skin flaps of some of the strain and pressure caused by the breast implants, acellular dermal matrixes (ADM) are increasingly used in this type of procedures. ADMs are derived from the skin of humans or animals, processed to an extent where their cellular components are completely removed, leaving only the extracellular scaffold, thus not inciting an immune response from the host. The ADM thus provides a scaffold, promoting integration of the patient's own connective tissue. In time the ADM will be repopulated and revascularized by the patient's own cells, essentially becoming an integrated part of the patients body. The ADM provides optimal definition of the breast borders, essentially allowing improved implant positioning as compared with a sub muscular coverage technique. If the circumstance of the breast reconstructions necessitates the placement of an expander implant, use of ADMs allows for a greater intraoperative expansion, and thus subsequently reduces the number of times the patients must attend the outpatient's clinic for expansion of the implant. Thus leading to a shorter time before the expander implant may be exchanged for a permanent implant. Furthermore, several studies have shown that use of ADM lowers the overall complication rate.

Several types of ADM are used in a breast reconstructive setting around the world. Strattice™ is a porcine derived ADM, and has been available in Europe and Denmark since late 2008. In order to find the best available ADM for use in a immediate breast reconstructive setting, both in terms of complication rates and patient satisfaction, it is crucial that new products are continuously evaluated. SurgiMend®, another type of ADM, was recently introduced on the Danish market. SurgiMend® ADM is derived from fetal bovine dermis, and recent studies show that the use of SurgiMend® ADM is associated with a low early complication rate. Furthermore, a recent study provided evidence that ADM derived from bovine have a higher mechanical stress tolerance when compared to porcine derived ADM at equivalent thickness.

Aim

The aim of the present study is to evaluate two types of ADM´s in an immediate breast reconstructive setting. The data from this study will possibly help to minimize complications and increase patient satisfaction by finding the optimal ADM for immediate breast reconstructions, thereby contributing to a faster recovery for women who undergo mastectomy and immediate breast reconstruction with implant and ADM.

Hypothesis

SurgiMend and Strattice™ provide equal results in regards to complication rates, patient reported outcome measures and aesthetic appearance in patients undergoing immediate breast reconstruction.

Methods

The project is conducted as a prospective randomized trial. Patients included in the study will be randomized to receive either Strattice™ or SurgiMend® ADM. Patients are allocated in a 1:1 ratio, with 30 patients receiving Strattice™ ADM and 30 patients receiving SurgiMend® ADM. The randomization is performed using a permuted block randomization. Randomization is blinded for the patients and the outcome assessor. Regardless of which type of ADM the patient is randomized to receive, the surgical procedure will be performed in the same way.

Patients included in the study will be asked to complete the BREAST-Q pre-reconstruction module before their breast reconstruction, and the BREAST-Q post-reconstruction module at 4 and 12 months after their breast reconstruction. The BREAST-Q is a patient reported outcome measure tool specifically designed and validated for use in breast reconstruction patients. The BREAST-Q modules consists of several scales, investigating the patients body image, satisfaction with breasts and satisfaction with care. The BREAST-Q modules are widely used and have been officially translated into the Danish language.

Participating patients will attend the same standard post-operative controls at 4 and 12 months after their breast reconstruction as non-participating patients undergoing immediate breast reconstruction. In addition to being examined by their operating surgeon at these controls, the patients' aesthetic result will be evaluated by one of the investigators using a breast reconstruction outcome scale, previously developed at Dept. of Plastic and Reconstructive Surgery, Aarhus University Hospital, Aarhus, Denmark. The scale consists of six questions evaluating the symmetry, feel, and aesthetic appearance of the reconstructed breasts.

Recruitment of participants

Patients seeking an immediate breast reconstruction are routinely seen in the Dept. of Plastic and Reconstructive Surgery patient clinic by both a consultant breast surgeon and a consultant plastic surgeon at the same time. If the breast and plastic surgeon deems the patient eligible for a primary breast reconstruction and the plastic surgeon evaluates the patient to be best suited with a breast reconstruction based on an implant and ADM, the patient will be offered a consultation with the clinical investigator for the project. If the plastic surgeon believes that a patient is a better candidate for another type of breast reconstructive procedure than implant and ADM, the patient will not be offered participation.

At the consultation with the investigator, or a well-instructed colleague, the patient will be given oral and written information about the research project. The patient will always be offered a period of at least 24 hours before deciding to give consent, but may also give her informed consent on site. Furthermore, the patient will be offered a second consultation, where the information about the project will be repeated and any questions regarding the research project she may have will be answered. The patient will also be encouraged to bring a family member or friend to the second meeting. The patient may at any time and without need of justification withdraw consent to participate, without affecting the present and/or future treatment of the patient.

Risks, side effects and disadvantages

As with all surgery, there is a risk of wound infection, blood clots and altered sensation in the operated area. This can lead to antibiotic treatment, or where appropriate, a second operation to stop bleeding or remove damaged tissue. These risks are, however, associated with the breast reconstruction itself, and not associated with participating in the current study.

Both types of ADM are well described in the medical literature, and both types of ADM have achieved good results compared to not using ADM in immediate breast reconstructions. The risks for the patients choosing to participate in the project are thus solely related to the breast reconstruction itself, and not to the participation in the current study.

Participating patients will have to spend approximately 10 minutes completing a questionnaire before the breast reconstruction. Additionally, the participating patients will be asked to complete another questionnaire (approximately 10 min) at 4 and 12 months after their breast reconstruction, as well as participate in an extra clinical examination at their routine follow-up examinations after 4 and 12 months. The extra examinations at the routine follow-up visits are expected to take approximately 15 min. per visit. While the questionnaire and the clinical follow-up may consume some of the patient's time, there are no risks associated with them.

Ethical considerations

It is expected that the number of women who choose an immediate breast reconstruction procedure will increase. Conducting studies that help bring down the complication rates for these types of surgery is of utmost importance, both for the individual patient undergoing the surgery and in a socio-economic setting.The proposed study will aid in finding the optimal method, both in terms of complication rate and patient reported outcome. All of the patients invited to participate in this study has been evaluated by experienced breast and plastic surgeons to be best suited with an immediate breast reconstruction with implant and ADM. The two types of ADMs evaluated in the study have shown good results in previous studies. As it is not expected that one of the tested ADMs is significantly better than the other, there is no predictable benefit for the individual patient in regards to participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been deemed eligible for an immediate breast reconstruction using implant and ADM by the responsible plastic and breast surgeon
* Patient is older than 18 years of age
* Patient understand enough Danish to comprehend the given information and to complete the study questionnaires

Exclusion Criteria:

* Current smokers (patients not having paused for a minimum of four weeks prior to surgery)
* Non-eligible patients, as assessed by operating surgeon
* High level of co-morbidity, as assessed by operating surgeon or anesthesiologist

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Complication Rate | 1 year from surgery
  The prevalence of complications to the BR.

SECONDARY OUTCOMES:
Patients reported satisfaction | 1 year
  Patient reported satisfaction as measured by the BREAST-Q.
Aesthetic result | 1 year
  The aesthetic outcome of the BR as evaluated by a clinician using a study specific breast reconstruction outcome scale.
Cost of Care | 1 year
  The total cost for the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tine E Damsgaard, MD, PHD, Principal Investigator — Plastic Surgery Research Unit, Dept. of Plastic Surgery, Aarhus University Hospital, Aarhus, Denmark
Locations (1):
- Dept. of Plastic Surgery, Aarhus University Hospital, Aarhus C, Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meijers-Heijboer H, van Geel B, van Putten WL, Henzen-Logmans SC, Seynaeve C, Menke-Pluymers MB, Bartels CC, Verhoog LC, van den Ouweland AM, Niermeijer MF, Brekelmans CT, Klijn JG. Breast cancer after prophylactic bilateral mastectomy in women with a BRCA1 or BRCA2 mutation. N Engl J Med. 2001 Jul 19;345(3):159-64. doi: 10.1056/NEJM200107193450301. PMID 11463009
- [Background] Skytte AB, Cruger D, Gerster M, Laenkholm AV, Lang C, Brondum-Nielsen K, Andersen MK, Sunde L, Kolvraa S, Gerdes AM. Breast cancer after bilateral risk-reducing mastectomy. Clin Genet. 2011 May;79(5):431-7. doi: 10.1111/j.1399-0004.2010.01604.x. Epub 2011 Jan 4. PMID 21199491
- [Background] Takami Y, Matsuda T, Yoshitake M, Hanumadass M, Walter RJ. Dispase/detergent treated dermal matrix as a dermal substitute. Burns. 1996 May;22(3):182-90. doi: 10.1016/0305-4179(95)00123-9. PMID 8726254
- [Background] Breuing KH, Warren SM. Immediate bilateral breast reconstruction with implants and inferolateral AlloDerm slings. Ann Plast Surg. 2005 Sep;55(3):232-9. doi: 10.1097/01.sap.0000168527.52472.3c. PMID 16106158
- [Background] Salzberg CA. Nonexpansive immediate breast reconstruction using human acellular tissue matrix graft (AlloDerm). Ann Plast Surg. 2006 Jul;57(1):1-5. doi: 10.1097/01.sap.0000214873.13102.9f. PMID 16799299
- [Background] Spear SL, Parikh PM, Reisin E, Menon NG. Acellular dermis-assisted breast reconstruction. Aesthetic Plast Surg. 2008 May;32(3):418-25. doi: 10.1007/s00266-008-9128-8. PMID 18338102
- [Background] Sbitany H, Sandeen SN, Amalfi AN, Davenport MS, Langstein HN. Acellular dermis-assisted prosthetic breast reconstruction versus complete submuscular coverage: a head-to-head comparison of outcomes. Plast Reconstr Surg. 2009 Dec;124(6):1735-1740. doi: 10.1097/PRS.0b013e3181bf803d. PMID 19952627
- [Background] Hanna KR, DeGeorge BR Jr, Mericli AF, Lin KY, Drake DB. Comparison study of two types of expander-based breast reconstruction: acellular dermal matrix-assisted versus total submuscular placement. Ann Plast Surg. 2013 Jan;70(1):10-5. doi: 10.1097/SAP.0b013e31822f6765. PMID 21862915
- [Background] Colwell AS, Damjanovic B, Zahedi B, Medford-Davis L, Hertl C, Austen WG Jr. Retrospective review of 331 consecutive immediate single-stage implant reconstructions with acellular dermal matrix: indications, complications, trends, and costs. Plast Reconstr Surg. 2011 Dec;128(6):1170-1178. doi: 10.1097/PRS.0b013e318230c2f6. PMID 22094736
- [Background] Endress R, Choi MS, Lee GK. Use of fetal bovine acellular dermal xenograft with tissue expansion for staged breast reconstruction. Ann Plast Surg. 2012 Apr;68(4):338-41. doi: 10.1097/SAP.0b013e31823b68d0. PMID 22421474
- [Background] Macadam SA, Lennox PA. Acellular dermal matrices: Use in reconstructive and aesthetic breast surgery. Can J Plast Surg. 2012 Summer;20(2):75-89. doi: 10.1177/229255031202000201. PMID 23730154
- [Background] Ho G, Nguyen TJ, Shahabi A, Hwang BH, Chan LS, Wong AK. A systematic review and meta-analysis of complications associated with acellular dermal matrix-assisted breast reconstruction. Ann Plast Surg. 2012 Apr;68(4):346-56. doi: 10.1097/SAP.0b013e31823f3cd9. PMID 22421476
- [Background] Breuing KH, Colwell AS. Inferolateral AlloDerm hammock for implant coverage in breast reconstruction. Ann Plast Surg. 2007 Sep;59(3):250-5. doi: 10.1097/SAP.0b013e31802f8426. PMID 17721209
- [Background] Bank J, Phillips NA, Park JE, Song DH. Economic analysis and review of the literature on implant-based breast reconstruction with and without the use of the acellular dermal matrix. Aesthetic Plast Surg. 2013 Dec;37(6):1194-201. doi: 10.1007/s00266-013-0213-2. Epub 2013 Oct 3. PMID 24091489
- [Background] Krishnan NM, Chatterjee A, Rosenkranz KM, Powell SG, Nigriny JF, Vidal DC. The cost effectiveness of acellular dermal matrix in expander-implant immediate breast reconstruction. J Plast Reconstr Aesthet Surg. 2014 Apr;67(4):468-76. doi: 10.1016/j.bjps.2013.12.035. Epub 2014 Jan 23. PMID 24508194
- [Background] Ohkuma R, Buretta KJ, Mohan R, Rosson GD, Rad AN. Initial experience with the use of foetal/neonatal bovine acellular dermal collagen matrix (SurgiMend) for tissue-expander breast reconstruction. J Plast Reconstr Aesthet Surg. 2013 Sep;66(9):1195-201. doi: 10.1016/j.bjps.2013.05.004. Epub 2013 Jun 13. PMID 23768943
- [Background] Butterfield JL. 440 Consecutive immediate, implant-based, single-surgeon breast reconstructions in 281 patients: a comparison of early outcomes and costs between SurgiMend fetal bovine and AlloDerm human cadaveric acellular dermal matrices. Plast Reconstr Surg. 2013 May;131(5):940-951. doi: 10.1097/PRS.0b013e3182865ab3. PMID 23629076
- [Background] Adelman DM, Selber JC, Butler CE. Bovine versus Porcine Acellular Dermal Matrix: A Comparison of Mechanical Properties. Plast Reconstr Surg Glob Open. 2014 Jun 6;2(5):e155. doi: 10.1097/GOX.0000000000000072. eCollection 2014 May. PMID 25289348
- [Background] Doig GS, Simpson F. Randomization and allocation concealment: a practical guide for researchers. J Crit Care. 2005 Jun;20(2):187-91; discussion 191-3. doi: 10.1016/j.jcrc.2005.04.005. PMID 16139163
- [Background] Pusic AL, Klassen AF, Scott AM, Klok JA, Cordeiro PG, Cano SJ. Development of a new patient-reported outcome measure for breast surgery: the BREAST-Q. Plast Reconstr Surg. 2009 Aug;124(2):345-353. doi: 10.1097/PRS.0b013e3181aee807. PMID 19644246